CLINICAL TRIAL: NCT03501186
Title: Effects of Backward Gait on Sand on Improving the Gait Parameters of Patients With Chronic Stroke: a Randomized Controlled Trial
Brief Title: Effects of Backward Gait on Sand on Improving the Gait Parameters of Patients With Chronic Stroke.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, faizan kashoo, PT, Faizan Kashoo, Master in physiotherapy, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Majmaah
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Chronic Stroke
Keywords: Backward walking, stroke, gait training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The treatment given by investigator unaware of allocation of patients and outcome variables measured by different investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): forward walking on leveled surface
  Interventions: Other: Backward walking on sand
- Group 2 (Active Comparator): forward walking on sand.
  Interventions: Other: Backward walking on sand
- Group 3 (Experimental): Backward walking on leveled surface
  Interventions: Other: Backward walking on sand
- Group 4 (Active Comparator): Backward walking on sand.
  Interventions: Other: Backward walking on sand

INTERVENTIONS:
Other: Backward walking on sand — the patient will be walking backwards on sand with therapist standing close to support in case of fall.
  Other Names: forward walking on sand

SUMMARY:
Gait training in stroke is a complex process of motor learning although restoring patients ability to walk would not prepare the individual with the challenges faced in the real environment. The aim is not simply walking in controlled environment, but to achieve dynamic walking. Dynamic walking is the ability of an individual to adjust to the changing surfaces and terrains. thereby returning to achieve active participation in the community. Hence, recovery of walking ability is the primary goal when planning treatment for patients with stroke.

ELIGIBILITY:
Inclusion criteria:

* Had experienced stroke for the first time.
* Unilateral involvement.
* Demonstrate motor stage 3 or 4 on Brunnstrom motor recovery.
* Able to walk 12 m with or without assistive devices.
* Medically stable.
* Able to follow simple commands.

Exclusion criteria:

* Patient exhibits comorbid disease other than stroke that may affect gait.
* Any conditions contra indicated to exercises
* Any other cardio-pulmonary or orthopedic disorders that affects walking ability of the participant.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01-12 (Actual); Primary Completion 2018-06-20 (Estimated); Study Completion 2018-07-21 (Estimated)

PRIMARY OUTCOMES:
Gait velocity (m/s) | 10-15 mins
  Measured by Stride Analyser
Cadence (Number of steps per min) | 10-15 mins
  Measured by stride Analyser
Stride length in meters | 10-15 mins
  Measured by stride Analyser
Gait cycle in seconds | 10-15 mins
  Measured by stride Analyser

SECONDARY OUTCOMES:
Barthel index | 45 Mins
  ADL

CONTACTS AND LOCATIONS:
Locations (1):
- King Khalid Hospital, Al Majma'ah, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Stroke Patients
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 months

REFERENCES:
- [Background] Makino M, Takami A, Oda A. Comparison of forward walking and backward walking in stroke hemiplegia patients focusing on the paretic side. J Phys Ther Sci. 2017 Feb;29(2):187-190. doi: 10.1589/jpts.29.187. Epub 2017 Feb 24. PMID 28265136
- [Background] Kim CY, Lee JS, Kim HD. Comparison of the Effect of Lateral and Backward Walking Training on Walking Function in Patients with Poststroke Hemiplegia: A Pilot Randomized Controlled Trial. Am J Phys Med Rehabil. 2017 Feb;96(2):61-67. doi: 10.1097/PHM.0000000000000541. PMID 27323323